CLINICAL TRIAL: NCT07003776
Title: Evaluation of Tumor Budding In Colorectal Adenocarcinoma
Status: Not yet recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Shaza Mostafa Galal Mostafa, demonstrator at pathology department, Sohag University
Other Study IDs: Soh-Med--25-5-2MS
Record Dates: First submitted 2025-05-26; First posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Colorectal Adenocarcinoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — 50 formalin fixed, paraffin embedded colorectal cancer tissue blocks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- paticipants: 50 archived Formalin-fixed Paraffin-embedded tissue blocks of Colorectal Carcinoma will be obtained and sectioned. From each block; Two tissue sections will be prepared, one tissue section will be stained by Hematoxylin and Eosin to detect tumor phenotype and depth of invasion. Other tissue section will be immunohistochemically stained by Pan-cytokeratin
  Interventions: Other: Biological: Immunohistochemical staining

INTERVENTIONS:
Other: Biological: Immunohistochemical staining — Staining of Colorectal Carcinoma tissue sections by monoclonal antibodies against Pan- cytokeratin by immunohistochemical procedures.

SUMMARY:
Colorectal cancer (CRC) is among the most prevalent cancers globally, with approximately one to two million new cases diagnosed each year. This makes CRC the third most common cancer and the fourth leading cause of cancer-related deaths, with 700,000 deaths per year, exceeded only by lung, liver and stomach cancers. CRC accounts for about 10% of all cancer diagnoses worldwide (Sung et al., 2021; Masetti et al., 2022) .

CRC affects different races and ethnicities at various age groups in distinct ways. Among patients younger than 50 years old, the proportion of CRC is nearly double for Black individuals (16%) compared to White individuals (9%) and Hispanic individuals (6%). In Egypt, CRC ranked the seventh among cancers, following lung, breast, prostate, liver, and bladder cancers (Mounir et al., 2022).

Tumor budding (TB) is characterized by the presence of individual tumor cells or small clusters of up to four cells at the invasive margin of a tumor. This histological feature, which indicates the separation of malignant cells from the main tumor mass, has intrigued pathologists since it was first identified in the 1950s (Giordano et al., 2024).

Evaluating TB is crucial for improving prognostic accuracy and informing treatment decisions. Tumors with high-grade TB exhibit a significantly lower 5-year Disease-Free Survival (DFS) rate compared to those with low-grade TB. High-grade TB is regarded as a negative prognostic factor and is associated with an increased risk of recurrence (Kyong Shin et al., 2023).

TB can be observed in conventional slides when prominent, but careful observation is necessary. A more thorough assessment of TB is more easily achieved if the neoplastic epithelium is highlighted using pan-cytokeratin immunostains (Mishra et al., 2022).

Pan-keratin (Pan-CK) antibodies are proteins derived from cytoskeletal intermediate filaments. These antibodies are a mixture designed to detect multiple low and high molecular weight keratins. Their primary purpose is to allow for the immunohistochemical identification of all epithelial cell types, regardless of their tissue of origin, using a single diagnostic tool.

In surgical pathology, Pan-CK antibodies are commonly used to confirm the epithelial origin of both neoplastic (tumorous) and non-neoplastic tissues, as well as to identify small metastases in lymph nodes. However, there are limitations to the assumption that Pan-CK antibodies will stain all epithelial tumors and that non-epithelial tissues will be "keratin negative." It has been reported that a diverse range of epithelial tumors can be Pan-CK negative, challenging the notion that these antibodies are universally applicable (Wick et al., 1986; Badzio, 2019).

Pan-CK can help diagnose disease like breast cancer, lung cancer, prostate cancer, and colorectal cancer. It is often used in conjunction with other antibodies for these specific cancers (Chu and Weiss, 2002).

ELIGIBILITY:
Inclusion Criteria:

* Specimens from patients with Colorectal Carcinoma. Tissue blocks with sufficient material. Specimens with sufficient clinical data.

Exclusion Criteria:

* Tissue blocks with insufficient, destroyed or necrotic material. Specimens with insufficient clinical data.

Ages: 20 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Archived Formalin-fixed, Paraffin-embedded tissue blocks belonged to patients suffered from colonic and/or rectal cancers. Patients were admitted to sohag university hospital and underwent colectomy and their colonic specimens were sent to Pathology Laboratory of the same hospital to ascertain diagnosis and tumor phenotype.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-05-03 (Estimated); Study Completion 2026-05-03 (Estimated)

PRIMARY OUTCOMES:
Evaluation of Tumor Budding in Colorectal Adenocarcinoma | 6 months
  Histological assessment and immunohistochemical highlighting of tumor Budding by Pan-CK.

SECONDARY OUTCOMES:
Correlation of Tumor Budding with clinicopathological parameters | 6 months
  Correlation between different grades of Tumor Budding in Colorectal Carcinoma cells and some clinical and pathological parameters as age, sex, tumor phenotype and nodal status.

REFERENCES:
- [Background] Wick MR, Cherwitz DL, McGlennen RC, Dehner LP. Adrenocortical carcinoma. An immunohistochemical comparison with renal cell carcinoma. Am J Pathol. 1986 Feb;122(2):343-52. PMID 2418689
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Background] Mounir, A., Hassan, M. A., Selim, M. A., and Mahmoud, I. A. (2022). Epidemiology of Colorectal Cancer, Incidence, Survival, and Risk Factors: Cairo University Center of Oncology and Nuclear Medicine Experience. The Egyptian Journal of Hospital Medicine, 89(2), 7061-7070. https://doi.org/10.21608/ejhm.2022.272513
- [Background] Masetti M, Fallani G, Ratti F, Ferrero A, Giuliante F, Cillo U, Guglielmi A, Ettorre GM, Torzilli G, Vincenti L, Ercolani G, Cipressi C, Lombardi R, Aldrighetti L, Jovine E. Minimally invasive treatment of colorectal liver metastases: does robotic surgery provide any technical advantages over laparoscopy? A multicenter analysis from the IGoMILS (Italian Group of Minimally Invasive Liver Surgery) registry. Updates Surg. 2022 Apr;74(2):535-545. doi: 10.1007/s13304-022-01245-1. Epub 2022 Jan 31. PMID 35099776
- [Background] Mishra, P. P., Madan, K., Biswas, S., Rao, A. C. K., Shetty, R., and Panda, P. (2022). Tumour budding in colorectal carcinoma: Association with other histopathological prognostic parameters. IP Archives of Cytology and Histopathology Research, 7(1), 26-31. https://doi.org/10.18231/j.achr.2022.006
- [Background] Kyong Shin J, Ah Park Y, Wook Huh J, Hyeon Yun S, Cheol Kim H, Yong Lee W, Hyung Kim S, Yun Ha S, Cho YB. Is High-Grade Tumor Budding an Independent Prognostic Factor in Stage II Colon Cancer? Dis Colon Rectum. 2023 Aug 1;66(8):e801-e808. doi: 10.1097/DCR.0000000000002345. Epub 2022 Apr 5. PMID 35394982
- [Background] Giordano PG, Diaz Zelaya AG, Aguilera Molina YY, Taboada Mostajo NO, Ajete Ramos Y, Ortega Garcia R, Peralta de Michelis E, Meneu Diaz JC. Clinico-pathological evaluation of tumor budding in the oncological progression of colorectal cancer. Med Clin (Barc). 2024 Aug 30;163(4):159-166. doi: 10.1016/j.medcli.2024.02.017. Epub 2024 May 1. English, Spanish. PMID 38697893
- [Background] Chu PG, Weiss LM. Keratin expression in human tissues and neoplasms. Histopathology. 2002 May;40(5):403-39. doi: 10.1046/j.1365-2559.2002.01387.x. PMID 12010363
- [Background] Badzio A, Czapiewski P, Gorczynski A, Szczepanska-Michalska K, Haybaeck J, Biernat W, Jassem J. Prognostic value of broad-spectrum keratin clones AE1/AE3 and CAM5.2 in small cell lung cancer patients undergoing pulmonary resection. Acta Biochim Pol. 2019 Feb 22;66(1):111-114. doi: 10.18388/abp.2018_2773. PMID 30793712